

# STUDY INFORMATION – Housing Outreach Project Collaborative (HOP-C) Participants

### Name of Study: Exiting Homelessness Intervention

**Responsible Investigators:** Sean Kidd 416-535-8501 ext. 36295, Centre for Addition and Mental Health (CAMH); Tyler Frederick 905-721-8668 ext. 5881, University of Ontario Institute of Technology; Kwame McKenzie, The Wellesley Institute, (416) 972-1010

**Purpose/description:** This project is being done to explore the impact of an intervention that supports youth in their transition away from homelessness for youth. The intervention and the study will last 6 months. Approximately 50 people will take part, randomly assigned to either case management only or a combination of case management, peer support and mental health support. You have been randomly assigned to the arm that includes case management, peer support and mental health support.

As part of this intervention you will:

- 1. Have access to a transitional caseworker. The caseworker's role is to provide you with support and advice in your transition away from homelessness. Examples of this may include support in the domains of housing, daily living, education/employment, and financial management, as well as assistance in accessing referrals.
- 2. Have access to a peer mentor. The peer mentor is a trained and supervised person who has previously experienced their own journey from homelessness to stable housing. The peer mentor's role is to provide support, advice and to organize social activities and hang outs. Peer mentors are available to meet with you one on one and/or during group outings and meeting. Activities organized by peer mentors will include arts and media projects, navigating activities at Sketch Arts, as well as monthly outings in the community involving movies, sports, board games and special events. The peer support worker will also be connecting with the wider team involved in this project e.g. case manager and researchers. You do not have to meet with the peer mentor, but we do ask that you meet with them a couple of times to see if you like it.
- 3. Have access to a weekly mental health and wellness group with a psychologist. These sessions will run weekly for 6 months and each session will last 90 minutes. It will be a place to discuss your experiences and challenges, and to learn some psychological techniques for improving your mental health and well-being. You do not have to attend the group sessions, but we ask that you try at least a couple to see if you like it.
- 4. Have access to family counselling sessions with a psychologist: You will have an opportunity to set up 3 family counselling sessions with a psychologist to address any family issues with members of your family you want to work on. You do not have to use these if you do not want to.

| ı | D۵ | rti | icina | nt's | Initials: |
|---|----|-----|-------|------|-----------|

5. Have access to individual psychotherapy with a psychologist. If you find that the other supports listed above are not helping, individual psychotherapy will be available for you to access. These sessions will provide you with support and strategies related to your mental health and well-being in a one to one setting. You do not have to use these sessions if you do not want to.

To explore the impact of the intervention as part of the study you will be expected to: Meet 2 times with a research assistant to complete surveys about your living circumstances, quality of life and mental health. One interview will be scheduled at the beginning and a final one at the end of the 6 months. The interviews will be approximately 1 hour in length. At the final interview you will be asked questions about what was more and less helpful about the intervention.

**Eligibility:** To take part in this study you must (i) be between 16 and 26 years of age, (ii) have been without a stable place to stay for 6 months total in your life (sleeping on the street, couch surfing, emergency shelters) (iii) been in stable housing for up to 12 months immediately prior to your first interview (i.e. your own apartment, room, or house where you or social assistance pays rent, transitional housing that you could stay at for a year or more, home of a family member or caregiver).

**Study Confidentiality:** Your identity will be kept private and confidential to the full extent provided by law. We will not identify you by name or in any other way that you could be recognized in any report that comes out of this study. However, there are some situations where we cannot guarantee your confidentiality. These are situations in which a participant was to tell us that he or she plans to commit suicide, kill another person, or tells us about a child that is being abused. In those situations we have a legal duty to act on that information and involve the appropriate service or authority to prevent harm.

The caseworkers, peer mentors, and psychologist are going to be interviewed about their role and experience in the intervention as well. They will not be asked questions specifically about their contacts with you – rather they will talk about their experience generally. They will also record the number of times that you meet with them, their feelings about the quality of the meetings, and their impressions about the main issues and challenges you are facing in your transition. This information will be pooled with other participants (e.g., averages) for analysis in the study. Any information about you that might arise in the interviews with the caseworker, peer, or psychologist will be kept confidential within the study to the full extent of the law as described above.

**Audio Recordings:** Audio recordings of your answers regarding the intervention at the second interview will be made. They will be destroyed within one month after they have been transcribed. Transcription is being done by the interviewer and a professional company that has signed a contract to keep the interviews and transcripts confidential.

| 1 | | | ., . | 1 | |
|---|-------|-------|----------|--------|----|
| | レコrtı | cipan | it'c In | ntiale | • |
| | | CIDAI | 11. 3 11 | пиан | ). |

**Ethics Review Board**: As part of continuing review of the research, your study records may be assessed on behalf of the Research Ethics Board. A person from the research ethics team may contact you (if your contact information is available) to ask you questions about the research study and your consent to participate. The person who looks at your file or contacts you must also keep your information private and confidential.

**Quality Assurance**: As part of the Research Services Quality Assurance Program, this study may be monitored and/or audited by a member of the Quality Assurance Team. Your research records and CAMH records may be reviewed during which confidentiality will be maintained as per CAMH policies and extent permitted by law.

**Risks:** We don't think that you will feel any physical discomfort due to taking part in this project. While psychological risk (feeling upset emotionally) is expected to be low, some parts of the surveys and interviews might be distressing for some people. We encourage anyone taking parting the project to discuss any distress with the research assistant. If needed, we can provide information about the supports that are available for people experiencing distress.

**Compensation:** You will receive \$25.00 for your time completing each of the 2 interviews, for a total of \$50 over the course of the study. You will also be given 2 transit tokens to cover travel costs to and from the interviews.

**Benefits:** No direct benefits from taking part in this intervention are guaranteed. Indirectly you might benefit from the knowledge that by taking part you could be helping to improve services for street-involved and formerly street-involved youth.

**Voluntary Participation:** Your participation in this intervention and study is voluntary. You can choose to stop taking part in the intervention and study at any time. If you decide to stop taking part during one of the interviews, you will get paid the full amount for taking part in that interview. If you stop taking part in the project before completing both interviews, we will use the interview material that you gave us up to the time you left unless you tell us that you don't want any of your information used. Your choice to not participate or your choice to withdraw will not affect any treatment needs that you might have at the Centre for Addiction and Mental Health, SKETCH, LOFT and Covenant House.

**Additional Information:** If you have questions about the study that are not answered in these Information Sheets, please ask them. Also, if you have questions in the future you may contact the study investigators at the telephone numbers given on the first page. Dr. Robert Levitan, Chair, Research Ethics Board, Centre for Addiction and Mental Health, can also be contacted to discuss your rights. Dr. Levitan may be reached at 416-535-8501, extension 34020

| Participant's | Initials: |
|---------------|-----------|

| AGREEMENT TO PARTICIPATE 1, | have read the Information Sheet for the study named 'The |
|---|---|
| Exiting Homelessness Intervention investigators understand the impartment in the impartment of the investigation of the impartment of the | n.' My role in this project is as a research volunteer to help the act of an intervention addressing the transition away from my, have all been answered. By signing this consent form I do a to voluntarily participate in the intervention and research erstand that the project will be completed exactly as it is er, a copy of which I have been given. |
| I understand I can stop taking par<br>to give any reason for ending my ր | t in the project at any time, without penalty, and do not have participation. |
| I consent to (please check the box | for each activity you are consenting to): |
| and my experiences in over the course of 6 r and will take about 1 h Being asked if I know a that person with an inf | ew and questionnaires about my experiences of homelessness the intervention. I would take part in these interviews 2 times months. Each of these interviews will be done in one session our to complete. Inother person who could take part in this study and providing formation sheet about the study. Is sistant to contact (write name |
| of person) at<br>get my new phone num<br>Assistant can't get in to<br>they have. When they<br>Assistant on a project l<br>Assistant will tell that<br>that he/she could be | (write phone # or email address) to mber or email address. This will be done only if the Research ouch with me by the phone number and/or email address that call this person they will identify themselves as a Research looking at housing and community participation. The Research person that they have lost touch with me and I had agreed contacted for up to date contact information. The Research them any information about me or about the nature of the |
| with a Research Assista | o share my goals for and level of participation in the program ant. They may share the general points of my case, but no nformation that I have asked to keep strictly confidential. |
| ☐ Being re-contacted three interview about potent | ough my contact information or case manager after my T2 tial participation in a follow-up interview to happen 6 months-leting my time in HOPC |
| | h Ethics Board, Centre for Addiction and Mental Health, may to discuss their rights. <b>Dr. Levitan can be reached at: 416-535-</b> |
| I agree to participate. | |
| Research Volunteer: Signature: | Person Obtaining Consent/Witness: Signature: |

| Date: | Date: |
|-----------------------------------------------|-------|
| Name: | Name: |
| I have been given a copy of this form to keep | |

### **STUDY INFORMATION – Transitional Case Management Participants**

## Name of Study: Exiting Homelessness Intervention

**Responsible Investigators:** Sean Kidd 416-535-8501 ext. 36295, Centre for Addition and Mental Health (CAMH); Tyler Frederick 905-721-8668 ext. 5881, University of Ontario Institute of Technology; Kwame McKenzie, The Wellesley Institute, (416) 972-1010

**Purpose/description:** This project is being done to explore the impact of an intervention that supports youth in their transition away from homelessness for youth. The intervention and the study will last 6 months. Approximately 50 people will take part, randomly assigned to either case management only or a combination of case management, peer support and mental health support. You have been randomly assigned to the case management arm of this study.

As part of this intervention you will:

Participant's Initials: \_\_\_\_\_

6. Have access to a transitional caseworker. The caseworker's role is to provide you with support and advice in your transition away from homelessness. Examples of this may include support in the domains of housing, daily living, education/employment, and financial management, as well as assistance in accessing referrals.

To explore the impact of the intervention as part of the study you will be expected to: Meet two times with a research assistant to complete surveys about your living circumstances, quality of life and mental health. One survey will be scheduled at the beginning and a final one at the end of the 6 months. At the final interview you will be asked questions about what was more and less helpful about the intervention. These contacts will be approximately 1 hour in length.

**Eligibility:** To take part in this study you must (i) be between 16 and 26 years of age, (ii) have been without a stable place to stay for 6 months total in your life (sleeping on the street, couch surfing, emergency shelters) (iii) been in stable housing for up to 12 months immediately prior to your first interview (your own apartment, room, or house where you or social assistance pays rent, transitional housing that you could stay at for a year or more, home of a family member or caregiver).

**Study Confidentiality:** Your identity will be kept private and confidential to the full extent provided by law. We will not identify you by name or in any other way that you could be recognized in any report that comes out of this study. However, there are some situations where we cannot guarantee your confidentiality. These are, for example, situations in which a participant was to tell us that he or she plans to commit suicide, kill another person, or tells us about a child that is being abused. In such situations we have a legal duty to act on that information and involve the appropriate service or authority to prevent harm.

The consuler are going to be intentity wed about their role and experience in the

ced questions specifically about their contacts with you

– rather they will talk about their experience generally. They will also record the number of times that you meet with them, their feelings about the quality of the meetings, and their impressions about the main issues and challenges you are facing in your transition. This information will be pooled with other participants (e.g., averages) for analysis in the study. Any information about you that might arise in the interviews with the caseworker, peer, or psychologist will be kept confidential within the study to the full extent of the law as described above.

**Audio Recordings**: Audio recordings of your answers regarding the intervention at the second interview will be made. The recordings will be destroyed within one month after they have been transcribed. Transcription is being done by the interviewer and a professional company that has signed a contract to keep the interviews and transcripts confidential.

**Ethics Review Board**: As part of continuing review of the research, your study records may be assessed on behalf of the Research Ethics Board. A person from the research ethics team may contact you (if your contact information is available) to ask you questions about the research study and your consent to participate. The person who looks at your file or contacts you must also keep your information private and confidential.

**Quality Assurance**: As part of the Research Services Quality Assurance Program, this study may be monitored and/or audited by a member of the Quality Assurance Team. Your research records and CAMH records may be reviewed during which confidentiality will be maintained as per CAMH policies and extent permitted by law.

**Risks:** We don't think that you will feel any physical discomfort due to taking part in this project. While psychological risk (feeling upset emotionally) is expected to be low, some parts of the surveys and interviews might be distressing for some people. We encourage anyone taking parting the project to discuss any distress with the research assistant. If needed, we can provide information about the supports that are available for people experiencing distress.

**Compensation:** You will receive \$25.00 for your time completing each of the 2 interviews, for a total of \$50 over the course of the study. You will also be given 2 transit tokens to cover travel costs to and from the interviews.

**Benefits:** No direct benefits from taking part in this intervention are guaranteed. Indirectly you might benefit from the knowledge that by taking part you could be helping to improve services for street-involved and formerly street-involved youth.

**Voluntary Participation:** Your participation in this intervention and study is voluntary. You can choose to stop taking part in the intervention and study at any time. If you decide to stop taking part during one of the interviews, you will get paid the full amount for taking part in that

| Participant's Initials: | project before completing both interviews, we will use |
|---|---|
| the interview material that you gave us | up to the time you left unless you tell us that you don't |

want any of your information used. Your choice to not participate or your choice to withdraw will not affect any treatment needs that you might have at the Centre for Addiction and Mental Health, SKETCH, LOFT and Covenant House.

**Additional Information:** If you have questions about the study that are not answered in these Information Sheets, please ask them. Also, if you have questions in the future you may contact the study investigators at the telephone numbers given on the first page. Dr. Robert Levitan, Chair, Research Ethics Board, Centre for Addiction and Mental Health, may be contacted by research subjects to discuss your rights. Dr. Levitan can be reached at: 416-535-8501, extension 34020.

Participant's Initials:

| AGREEMENT TO PARTICIPATI | |
|---|---|
| have read the Information Sheet for the study named 'The exiting Homelessness Intervention.' My role in this project is as a research volunteer to help the investigators understand the impact of an intervention addressing the transition away from somelessness. My questions, if any, have all been answered. By signing this consent form I do not waive any of my rights. I agree to voluntarily participate in the intervention and research and give my consent freely. I understand that the project will be completed exactly as it is described in the Information Letter, a copy of which I have been given. | |
| I understand I can stop taking<br>to give any reason for ending | part in the project at any time, without penalty, and do not have my participation. |
| I consent to (please check the | e box for each activity you are consenting to): |
| and my experience over the course of and will take about Being asked if I know that person with a Allow the Research of person) at get my new phone Assistant can't get they have. When Assistant on a project Assistant will tell that he/she could Assistant will not research project. Allow my casework with a Research Assistant on a project. Being re-contacted interview about points. | erview and questionnaires about my experiences of homelessnesses in the intervention. I would take part in these interviews 2 time f 6 months. Each of these interviews will be done in one session t 1 hour to complete. ow another person who could take part in this study and providing n information sheet about the study. h Assistant to contact |
| , | earch Ethics Board, Centre for Addiction and Mental Health, may jects to discuss their rights. <b>Dr. Levitan can be reached at: 416-535-</b> |
| I agree to participate. | |
| Research Volunteer: Signature: | Person Obtaining Consent/Witness: Signature: |

| Date: | Date: |
|------------------------------------------------|-------|
| Name: | Name: |
| I have been given a copy of this form to keep. | |

#### STUDY INFORMATION – Toronto HOP-C Intervention Team Member

Name of Study: Exiting Homelessness Intervention

**Responsible Investigators:** Sean Kidd 416-535-8501 ext. 36295, Centre for Addition and Mental Health (CAMH); Christopher Mushquash (807) 343-8239; Tyler Frederick 905-721-8668 ext. 5881, University of Ontario Institute of Technology; Kwame McKenzie, The Wellesley Institute, (416) 972-1010

**Purpose:** This project is being done to explore the effectiveness of an intervention that supports youth in their transition away from homelessness. The intervention and the study will last 6 months, comparing the outcomes of youth engaged in case management alone versus the full HOP-C intervention. To explore the impact of the intervention as part of the study you will be expected to:

1. Participate in an interview with a researcher at the end of the 6 month study period regarding your experience and recommendations as a member of the intervention team (as a caseworker, psychologist, facilitator, peer worker, agency lead, or other role). This interview will be scheduled during work hours and at your convenience.

**Eligibility:** To take part in this study you must be a member of the intervention team as a caseworker, psychologist, facilitator, peer worker, agency lead, or other team role.

**Study Confidentiality:** Your identity will be kept private and confidential to the full extent provided by law. We will not identify you by name, only by general role, in any report that comes out of this study.

**Audio Recordings:** Audio recordings will be made of your interview. They will be destroyed within one month after they have been transcribed. Transcription is being done by a professional company that has signed a contract to keep the interviews and transcripts confidential.

**Ethics Review Board**: As part of continuing review of the research, your study records may be assessed on behalf of the Research Ethics Board. A person from the research ethics team may contact you (if your contact information is available) to ask you questions about the research study and your consent to participate. The person who looks at your file or contacts you must also keep your information private and confidential.

| Participant's Initials: |
|-------------------------|
|-------------------------|

**Quality Assurance**: As part of the Research Services Quality Assurance Program, this study may be monitored and/or audited by a member of the Quality Assurance Team. Your research records and CAMH records may be reviewed during which confidentiality will be maintained as per CAMH policies and extent permitted by law.

**Risks:** We don't expect there to be any risks associated with participation in this research.

**Compensation:** There will be no compensation for your participation in the research outside of the enumeration being received as part of your role in the intervention.

**Benefits:** No direct benefits are anticipated aside from some possible indirect benefit of being a part of this effort to better support marginalized young people.

**Voluntary Participation:** Your participation in this research is voluntary. You can choose to stop participating in the research at any time. If you stop taking part in the project before the completion of all interviews we will use the material that we have collected unless you tell us that you don't want any of your information used.

**Additional Information:** If you have questions about the study that are not answered in these Information Sheets, please ask them. Also, if you have questions in the future you may contact the study investigators at the telephone numbers given on the first page. Dr. Robert Levitan, Chair, Research Ethics Board, Centre for Addiction and Mental Health, may be contacted by research subjects to discuss their rights. Dr. Levitan can be reached at: 416-535-8501, extension 34020.

| Participant's Initials: |
|-------------------------|

| AGREEMENT TO PARTICIPATE | |
|---|---|
| ,, have read the Information Sheet for the study named 'The Exiting Homelessness Intervention.' My role in this aspect of the project is as a research volunteer based on my involvement as a member of the intervention team. My participation as a research volunteer will help the investigators understand the process of implementing the intervention and how features of the intervention shaped outcomes. My questions, if any, have all been answered. By signing this consent form I do not waive any of my rights. I agree to voluntarily participate in the research and give my consent freely. I understand that the project will be completed exactly as it is described in the Information Letter, a copy of which I have been given. | |
| I understand I can stop taking part in the research a have to give any reason for ending my participation | |
| I consent to (please check the box for each activity | you are consenting to): |
| ☐ Completing an interview about my expe | rience as a member of the research team |
| Dr. Robert Levitan, Chair, Research Ethics Board, Ce be contacted by research subjects to discuss their ri <b>8501</b> , extension <b>34020</b> . | - |
| I agree to participate. | |
| Research Volunteer: | Person Obtaining Consent/Witness: |
| Signature: | Signature: |
| Date: | Date: |
| Name: Name: | |
| I have been given a copy of this form to keep. | |

## STUDY INFORMATION – LPRF Thunder Bay HOP-C North Team Member

Name of Study: Exiting Homelessness Intervention

**Responsible Investigators:** Sean Kidd 416-535-8501 ext. 36295, Centre for Addition and Mental Health (CAMH); Christopher Mushquash (807) 343-8239; Tyler Frederick 905-721-8668 ext. 5881, University of Ontario Institute of Technology; Kwame McKenzie, The Wellesley Institute, (416) 972-1010

**Purpose:** This project is being done to better understand the relevance and outcomes of an intervention designed to support formerly homeless Indigenous youth successfully transition into housing and stability in their communities. As a part of this effort we are asking that you:

2. Participate in an interview with a researcher at the end of the 6 month study period regarding your experience and recommendations as a member of the intervention team (as a caseworker, psychologist, facilitator, peer worker, agency lead, or other role). This interview will be scheduled during work hours and at your convenience.

**Eligibility:** To take part in this study you must be a member of the intervention team as a caseworker, psychologist, facilitator, peer worker, agency lead, or other team role.

**Study Confidentiality:** Your identity will be kept private and confidential to the full extent provided by law. We will not identify you by name, only by general role, in any report that comes out of this study.

**Audio Recordings:** Audio recordings will be made of your interview. They will be destroyed within one month after they have been transcribed. Transcription is being done by a professional company that has signed a contract to keep the interviews and transcripts confidential.

**Ethics Review Board**: As part of continuing review of the research, your study records may be assessed on behalf of the Research Ethics Board. A person from the research ethics team may contact you (if your contact information is available) to ask you questions about the research study and your consent to participate. The person who looks at your file or contacts you must also keep your information private and confidential.

| Participant's Initials: |
|---------------------------------------------------|
| Quality Assurance: INSERT LOCALLY RELEVANT CONTEN |

**Risks:** We don't expect there to be any risks associated with participation in this research.

**Compensation:** There will be no compensation for your participation in the research outside of the enumeration being received as part of your role in the intervention.

**Benefits:** No direct benefits are anticipated aside from some possible indirect benefit of being a part of this effort to better support marginalized young people.

**Voluntary Participation:** Your participation in this research is voluntary. You can choose to stop participating in the research at any time. If you stop taking part in the project before the completion of all interviews we will use the material that we have collected unless you tell us that you don't want any of your information used.

**Additional Information:** If you have questions about the study that are not answered in these Information Sheets, please ask them. Also, if you have questions in the future you may contact the study investigators at the telephone numbers given on the first page. INSERT RELEVANT REB CHAIR CONTACT INFO

| Participant's | Initials: |
|---------------|-----------|

| AGREEMENT TO PARTICIPATE | |
|---|---|
| I,, have read the Inf<br>Exiting Homelessness Intervention.' My role in this<br>volunteer based on my involvement as a member of<br>a research volunteer will help the investigators und<br>intervention and how features of the intervention<br>all been answered. By signing this consent form I devoluntarily participate in the research and give my<br>will be completed exactly as it is described in the Influence given. | aspect of the project is as a research of the intervention team. My participation as derstand the process of implementing the shaped outcomes. My questions, if any, have o not waive any of my rights. I agree to consent freely. I understand that the project |
| I understand I can stop taking part in the research have to give any reason for ending my participation | |
| I consent to (please check the box for each activity | you are consenting to): |
| ☐ Completing an interview about my expe | erience as a member of the research team |
| LOCALLY RELEVANT CONTACT INTO | |
| I agree to participate. | |
| Research Volunteer: Signature: | Person Obtaining Consent/Witness: Signature: |
| Date: | Date: |
| Name: | Name: |
| I have been given a copy of this form to keep. | |